CLINICAL TRIAL: NCT00190307
Title: Strategy for Managing Antiplatelet Therapy in the Perioperative Period of Non Coronary Surgery
Brief Title: STRATAGEM: Strategy for Managing Antiplatelet Therapy in the Perioperative Period of Non Coronary Surgery
Acronym: STRATAGEM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Sanofi-Synthelabo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: P030440
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2011-09-21 (Estimated); Status verified 2005-09

CONDITIONS: Thrombosis
Keywords: Long term antiplatelet therapy; Scheduled surgery
MeSH Terms: conditions — Thrombosis | interventions — Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Aspirin:KARDEGIC
  Interventions: Drug: aspirin 75 mg/day

INTERVENTIONS:
Drug: aspirin 75 mg/day — aspirin 75 mg/day

SUMMARY:
The STRATAGEM trial is an investigator-driven French nationwide multicenter, randomized, double-blind, placebo-controlled trial comparing perioperative low-dose aspirin therapy versus placebo in the perioperative period in patients with documented symptomatic stable atherothrombotic disease taking antiplatelet therapy and undergoing non-coronary surgery.

DETAILED DESCRIPTION:
There is little evidence to guide antiplatelet therapy in patients at high risk of atherothrombotic events undergoing non cardiac surgery. Specifically, it is uncertain whether patients currently on antiplatelet therapy should continue or not continue treatment in the perioperative period.

Aim: To determine an evidence-based strategy for managing antiplatelet therapy in the perioperative period.

Methods: The STRATAGEM trial is an investigator-driven French nationwide multicenter, randomized, double-blind, placebo-controlled trial comparing perioperative low-dose aspirin therapy versus placebo in the perioperative period in patients with documented symptomatic stable atherothrombotic disease taking antiplatelet therapy and undergoing non-coronary surgery. The trial will involve 1500 patients at high risk of atherothrombosis, currently receiving long-term antiplatelet therapy and scheduled for non-coronary surgery in 50 centers. Ten days prior to surgery, patients will discontinue antiplatelet therapy and be randomly assigned to either 75 mg of aspirin or matching placebo for 10 days up to the surgical procedure. Usual therapy will be resumed after surgery according to local practice.

The main outcome measure will be a composite endpoint at day 30 reflecting serious perioperative complications, i.e. total mortality, severe ischemic events (ischemic stroke, non-fatal myocardial infarction [MI], acute limb ischemia, clinical deep venous thrombosis) and/or major hemorrhage (life-threatening bleeding or conducive to revision, or redo surgery, cerebral hemorrhage, intra- or retroperitoneal bleeding, bleeding resulting in the transfusion of more than 2 units of packed red blood cells). The hypothesis to be tested is that low-dose aspirin is associated with a net clinical benefit compared to placebo in the prevention of severe perioperative thrombotic and hemorrhagic complications.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Patients over eighteen years of age
* Patients treated with oral antiplatelet agents for secondary prevention (i.e. established and symptomatic cardiovascular disease):

  * regardless of the reason (coronary artery disease, stroke or TIA [transient ischemic attack], peripheral arterial disease)
  * regardless of the antiplatelet agent (aspirin, clopidogrel, ticlopidine, dipyridamole).
* Patients scheduled for intermediate or high-risk surgery, including but not limited to:

  * any long procedure associated with hemodynamic variations or major blood loss
  * valvular surgery
  * thoracic surgery
  * orthopedic surgery
  * general (intraperitoneal) surgery
  * urological surgery
  * vascular surgery
  * ear, nose, and throat (ENT) cancerology-related surgery.

Exclusion Criteria:

* Coronary bypass grafting surgery
* History of thrombocytopenia or allergy to heparin
* Arterial stent placement within the previous 30 days
* Active bleeding
* Formal contraindication to the use of anticoagulants and aspirin
* Recent acute coronary syndrome
* Ophthalmological surgery (posterior chamber)
* Neurosurgery
* Emergency surgery
* Thrombotic or bleeding risk deemed unacceptable by the surgical and anesthetic team
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 293 (Actual)
Dates: Start 2005-06; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Consisting of major thromboembolic events listed in the following table with their respective weights. | A composite criterion measured at Day 30
  The score allocated to each patient is the weight of the event (zero if no event has occurred). For the patients having experienced more than one event, the score attributed is the "heaviest" weight among the events he has undergone.

CONTACTS AND LOCATIONS:
Overall Officials: Jean Mantz, MD, Principal Investigator — Hôpital Beaujon, Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Beaujon, Clichy, France

REFERENCES:
- [Result] Mantz J, Samama CM, Tubach F, Devereaux PJ, Collet JP, Albaladejo P, Cholley B, Nizard R, Barre J, Piriou V, Poirier N, Mignon A, Schlumberger S, Longrois D, Aubrun F, Farese ME, Ravaud P, Steg PG; Stratagem Study Group. Impact of preoperative maintenance or interruption of aspirin on thrombotic and bleeding events after elective non-cardiac surgery: the multicentre, randomized, blinded, placebo-controlled, STRATAGEM trial. Br J Anaesth. 2011 Dec;107(6):899-910. doi: 10.1093/bja/aer274. Epub 2011 Aug 27. PMID 21873632